CLINICAL TRIAL: NCT03187496
Title: A Non-Randomized, Multiple-Dose, Open-Label, Single Sequence Study to Evaluate the Effect of Concomitant Administration of EDP-305 on the Pharmacokinetics and Safety of Midazolam, Caffeine, and Rosuvastatin in Healthy Human Volunteers
Brief Title: Drug-drug Interaction Study Between EDP-305, Midazolam, Caffeine and Rosuvastatin in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EDP 305-004
Record Dates: First submitted 2017-06-01; First posted 2017-06-15 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: NASH
Keywords: drug-drug interaction
MeSH Terms: interventions — Midazolam; Caffeine; Rosuvastatin Calcium; EDP-305

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Midazolam; Drug: Caffeine; Drug: Rosuvastatin; Drug: EDP-305

INTERVENTIONS:
Drug: Midazolam — Each subject will receive midazolam on Days 1 and 12.
Drug: Caffeine — Each subject will receive caffeine on Days 1 and 12.
Drug: Rosuvastatin — Each subject will receive rosuvastatin on Days 2 and 13.
Drug: EDP-305 — Each subject will receive EDP-305 on Days 5 through 15.

SUMMARY:
A non-randomized, multiple-dose, open-label, single sequence study to evaluate effect of concomitant administration of EDP-305 on the pharmacokinetics and safety of midazolam, caffeine, and rosuvastatin in healthy human volunteers.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 55 years, inclusive.
* Female subjects must be of non-childbearing potential.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease.
* Pregnant or nursing females.
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
* A positive urine drug screen at screening or Day -1.
* Current tobacco smokers or use of tobacco within 3 months prior to screening.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy).
* History of regular alcohol consumption.
* Participation in a clinical trial within 30 days prior to the first dose of study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Cmax of midazolam, caffeine, and rosuvastatin with and without the coadministration of EDP-305. | Up to 17 Days
AUC of midazolam, caffeine, and rosuvastatin with and without the coadministration of EDP-305. | Up to 17 days

SECONDARY OUTCOMES:
Cmax of 1'-hydroxymidazolam, paraxanthine and N-desmethyl-rosuvastatin with and without the coadministration of EDP-305. | Up to 17 days
AUC of 1'-hydroxymidazolam, paraxanthine and N-desmethyl-rosuvastatin with and without the coadministration of EDP-305. | Up to 17 days
Tmax of midazolam, 1'-hydroxymidazolam, caffeine, paraxanthine, rosuvastatin and N-desmethyl-rosuvastatin with and without the coadministration of EDP-305. | Up to 17 days
t1/2 of midazolam, 1'-hydroxymidazolam, caffeine, paraxanthine, rosuvastatin and N-desmethyl-rosuvastatin with and without the coadministration of EDP-305. | Up to 17 days
CL/F of midazolam, caffeine and rosuvastatin with and without the coadministration of EDP-305. | Up to 17 days
Vd/F of midazolam, 1'-hydroxymidazolam, caffeine, paraxanthine, rosuvastatin and N-desmethyl-rosuvastatin with and without the coadministration of EDP-305. | Up to 17 days
AUC ratios for 1'-hydroxymidazolam/midazolam, paraxanthine/caffeine, and N-desmethyl-rosuvastatin/rosuvastatin. | Up to 17 days
Safety measured by adverse events, physical exams, vital signs, 12-lead electrocardiograms (ECGs) and clinical lab results (including chemistry, hematology, and urinalysis). | Up to 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Dickerson, MD, Principal Investigator — Pharmaceutical Research Associates
Locations (1):
- Pharmaceutical Research Associates, Inc.,, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
When the clinical study report has been submitted to the appropriate Regulatory authorities, a lay person summary will be provided to all study subjects by mail or email.